CLINICAL TRIAL: NCT03599310
Title: Effects of a Structured Advance Care Planning Guide Among Patients With Advanced Illness in Hospital Care Settings: a Stepped-wedge Cluster Randomised Controlled Trial
Brief Title: Effects of a Structured Advance Care Planning Guide Among Patients With Advanced Illness in Hospital Care Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Food and Health Bureau, Hong Kong (Other Government)
Collaborators: Yan Chai Hospital (Other)
Responsible Party: Principal Investigator, Dr. Helen YL Chan, Associate Professor, Chinese University of Hong Kong
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 14152631
Record Dates: First submitted 2018-07-15; First posted 2018-07-26 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: End Stage Disease
Keywords: Advance care planning; Communication; Nurse; End-of-life
MeSH Terms: conditions — Communication; Death | interventions — Advance Care Planning

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Advance care planning (Experimental): The intervention is a facilitator-based ACP process with a structured guide as a communication tool to aid the interventionists in broaching end-of-life care issues and eliciting patients' values and preferences in a consistent manner.
  Interventions: Behavioral: Advance care planning
- Usual care (Placebo Comparator): A leaflet covering the concept of ACP and advance directives (AD), purposes and potential benefits will be distributed to all participants as part of usual information support to standardize the information provided. The health care team will encourage patients to discuss the matters with their family carers and/or significant others.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Advance care planning — The ACP guide is adapted from the Serious Illness Communication Guide and a culturally-sensitive ACP programme developed in the local context. The trained ACP facilitators will initiate the conversation by introducing the concepts of ACP with the support of the guide and assessing the patient's illness understanding and readiness to think about end-of-life care issues.
  Arms: Advance care planning
Behavioral: Usual care — In the current practice, patients will have to take the initiative themselves if they would like to discuss their end-of-life care or make an advance directive.
  Arms: Usual care

SUMMARY:
Objective: To examine the effects of a structured advance care planning (ACP) guide among patients with advanced illness in hospital care setting.

Methods: This is a 24-month stepped-wedge cluster randomised controlled trial to be conducted in the Department of Medicine in an acute hospital. Patients are eligible to the study if they are aged 18 or over, are communicable, and meet the indicators of health deterioration or advanced condition in the Supportive and Palliative Care Indicators Tool (SPICT). Ward nurses will be trained to be interventionists to conduct ACP by means of a structured ACP guide. The guide is adapted from a culturally sensitive ACP programme developed in the local context with reference to the format of the Serious Illness Communication Guide, which is an evidence-based best practice in end-of-life care communication to support the ACP process.

Main outcome measures: Data will be collected at baseline (T0), one week (T1), three months (T2) and six months (T3) after intervention. The primary study outcome is the documentation of ACP discussion in medical records and completion of advance directives. Secondary outcomes are communicating end-of-life care preferences with family carers, quality of life and concordance of care preferences and treatment provided.

DETAILED DESCRIPTION:
Advance care planning (ACP) is defined as a communication process among patients, their family members and healthcare providers about end-of-life care, before the patients lose their capacity to decide for themselves. The main purpose of this study is to embed ACP into the usual care process in acute hospital setting through building staff capacity to conduct ACP. This will be a 24-month stepped-wedge cluster randomised controlled trial, with randomization built into the phasing of intervention implementation. This crossover design enables all study venues sequentially switched from control to experimental. This study will be conducted in all eight wards of the medical department of an 800-bed acute hospital. The ACP in this study is a facilitator-based intervention with a structured communication guide as a tool to aid the interventionists in broaching end-of-life care issues and eliciting patients' values and preferences in a consistent manner. The primary study outcome is the documentation of ACP discussion in medical records. Secondary outcomes are communicating end-of-life care preferences with family carers, quality of life and concordance of care preferences and treatment provided. Data collection will be conducted at baseline, one week, three months and six months after intervention.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or over;
* meet either two general indicators of health deterioration or one clinical indicator of an advanced illness condition in the Supportive and Palliative Care Indicators Tool (SPICT); and
* able to communicate in Cantonese.

Exclusion Criteria:

* mentally incompetent or unable to communicate;
* receiving psychiatric treatment; or
* have been referred to the palliative care service at the time of recruitment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Documentation | 3 months
  Documentation of ACP discussion in medical record

SECONDARY OUTCOMES:
Family communication | 3 months
  Communication of end-of-life care preferences with family members
Self perceived quality-of-life of patients | 3 months
  Quality-of-life concerns at the end of life (QOLC-E)
Concordance of care | 6 months
  Concordance of care preferences and actual

CONTACTS AND LOCATIONS:
Overall Officials: Helen Y Chan, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Yan Chai Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Health conditions only